CLINICAL TRIAL: NCT01484561
Title: A Phase 1, Randomized, Placebo-Controlled, Two-Period, Fixed Sequence Study To Evaluate The Effect Of CP-690,550 On Measured Glomerular Filtration Rate In Patients With Active Rheumatoid Arthritis
Brief Title: A Study To Evaluate The Effect Of CP-690,550 On Measures Of Kidney Function In Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: A3921152
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Phase 1
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence 1 (Active Comparator)
  Interventions: Drug: CP-690,550 or Placebo
- Sequence 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CP-690,550 or Placebo — CP-690,550 10 mg twice a day (BID) orally or placebo BID orally, approximately 72 days
  Arms: Sequence 1
Drug: Placebo — Placebo BID orally, approximately 72 days
  Arms: Sequence 2

SUMMARY:
The purpose of study is to explore the effect of CP-690,550 (Tofacitinib) on measures of kidney function in patients with active rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* The patient must meet the American College of Rheumatology (ACR) classification criteria for the diagnosis of rheumatoid arthritis by satisfying at least four of the seven criteria.
* The patient must have active disease at both Screening and predose on Day 1 of Period 1.
* Patient must have had an inadequate response to at least one disease-modifying antirheumatic drug (DMARD), non-biologic or biologic, due to ineffectiveness or intolerance.

Exclusion Criteria:

* Pregnant or lactating women
* Serious medical conditions that would make treatment with CP-690,550 potentially unsafe.
* A patient who has a history of asthma, multiple allergies or severe allergy (eg, anaphylaxis) to any substance. In particular, a history of allergy to iodine, povidone-iodine, iohexol or other iodinated contrast media.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (5):
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Tacoma, Washington
- Pfizer Investigational Site, Prague, Czechia
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Würzburg
- Pfizer Investigational Site, Mérida, Yucatán, Mexico
- Poland (4):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Russia (3):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Petrozavodsk
  - Pfizer Investigational Site, Saint Petersburg
- Pfizer Investigational Site, Seoul, South Korea
- Spain (4):
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Barakaldo, Vizcaya
  - Pfizer Investigational Site, Bilbao, Vizcaya
  - Pfizer Investigational Site, A Coruña

REFERENCES:
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Kremer JM, Kivitz AJ, Simon-Campos JA, Nasonov EL, Tony HP, Lee SK, Vlahos B, Hammond C, Bukowski J, Li H, Schulman SL, Raber S, Zuckerman A, Isaacs JD. Evaluation of the effect of tofacitinib on measured glomerular filtration rate in patients with active rheumatoid arthritis: results from a randomised controlled trial. Arthritis Res Ther. 2015 Apr 6;17(1):95. doi: 10.1186/s13075-015-0612-7. PMID 25889308
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921152&StudyName=A%20Study%20To%20Evaluate%20The%20Effect%20Of%20CP-690%2C550%20On%20Measures%20Of%20Kidney%20Function%20In%20Patients%20With%20Active%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550/Placebo: Participants received CP-690,550 10 milligram (mg) tablets twice daily (BID) orally for 43 days (up to a maximum of 50 days) in Period 1 (43 days) followed immediately by placebo BID orally for 29 days (up to a maximum of 36 days) in Period 2
- Placebo/Placebo: Participants received matching placebo tablets orally for 43 days (up to a maximum of 50 days) in Period 1 immediately followed by matching placebo tablets orally for 29 days (up to a maximum of 36 days)
Period: Overall Study
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Started | 97 | 51
Completed | 88 | 45
Not Completed | 9 | 6
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Other | 1 | 1
Not completed — Adverse Event | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550/Placebo | Placebo/Placebo | Total
Number analyzed (Participants) | 97 | 51 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.7) | 47.3 (11.8) | 50.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 36 | 111
  Male | 22 | 15 | 37

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric (Geo) Mean-Fold Change at End of Period 1 From Baseline in Measured Glomerular Filtration Rate (mGFR)
Description: Glomerular filtration rate (GFR) is an index of kidney function. GFR describes the flow rate of filtered fluid through the kidney. GFR can be measured directly or estimated using established formulas. mGFR was determined using iohexol serum clearance using compartmental modeling of the iohexol serum concentration-time data. mGFR values were normalized to 1.73 meters squared (m^2) body surface area. A normal GFR is greater than (>)90 milliliters per minute (mL/min), although children and older people usually have a lower GFR. Lower values indicate poor kidney function. A GFR <15 mL/min is consistent with kidney failure. Baseline was defined as the mean of the values obtained at Run-in and on predose in Period 1/Day 1.
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of the test article (CP-690,550 or placebo). Observed Case (OC): missing data were not imputed. One participant was excluded (took wrong treatment) from FAS analysis of change at end of Period 1 from baseline in mGFR.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 91 | 46
fold change | 0.91 [0.88 to 0.95] | 0.99 [0.94 to 1.04]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold Change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 0.92, 90% CI 2-sided [0.86 to 0.98] — Analysis of covariance (ANCOVA) with change in logarithmic mGFR from baseline as dependent variable, treatment and logarithmic baseline as covariate

2. Secondary Outcome: Adjusted Geometric Mean-Fold Change at the End of Period 2 From Baseline in mGFR
Description: mGFR was determined using iohexol serum clearance using compartmental modeling of the iohexol serum concentration-time data. mGFR values were normalized to 1.73 m^2 body surface area. Baseline was defined as the mean of the values obtained at Run-in and on predose in Period 1/Day 1.
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS OC; three participants were excluded (took wrong treatment) from the FAS analysis of change at end of Period 2 from baseline in mGFR.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 86 | 45
fold change | 0.96 [0.92 to 1.00] | 0.92 [0.87 to 0.97]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 1.04, 90% CI 2-sided [0.97 to 1.11] — ANCOVA with change in logarithmic mGFR from baseline as dependent variable, treatment and logarithmic baseline as covariate

3. Secondary Outcome: Adjusted Geometric Mean-Fold Change at End of Period 2 From End of Period 1 in mGFR
Description: mGFR was determined using iohexol serum clearance using compartmental modeling of the iohexol serum concentration-time data. mGFR values were normalized to 1.73 m^2 body surface area.
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS OC; three participants were excluded (took wrong treatment) from the FAS analysis of change at end of Period 2 from end of Period 1 in mGFR.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 86 | 45
fold change | 1.03 [0.99 to 1.07] | 0.95 [0.90 to 0.99]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 1.09, 90% CI 2-sided [1.02 to 1.16] — ANCOVA with change in logarithmic mGFR from Period 2 baseline/the end of Period 1 as dependent variable, treatment and logarithmic Period 2 baseline/the end of Period 1 as covariate

4. Secondary Outcome: Adjusted Geometric Mean-Fold Change at End of Period 1 From Baseline in Estimated Glomerular Filtration Rate (eGFR) Using Modified Diet in Renal Disease (MDRD)
Description: eGFR was calculated using the MDRD equation and normalized to 1.73 m^2 body surface area. Baseline was defined as the mean of the values obtained at Screening and on predose in Period 1/Day 1.
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS (OC); one participant was excluded (took wrong treatment) from the FAS analysis of change at end of Period 1 from baseline in eGFR (MDRD).
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 92 | 46
fold change | 0.96 [0.94 to 0.97] | 1.01 [0.99 to 1.04]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 0.94, 90% CI 2-sided [0.91 to 0.97] — ANCOVA with change in logarithmic eGFR (MDRD) from baseline as dependent variable, treatment and logarithmic baseline as covariate

5. Secondary Outcome: Adjusted Geometric Mean-Fold Change at End of Period 2 From Baseline in eGFR Using MDRD
Description: eGFR was calculated using the MDRD equation with eGFR values normalized to 1.73 m^2 body surface area. Baseline was defined as the mean of the values obtained at Screening and on predose in Period 1/Day 1.
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS OC; three participants were excluded (took wrong treatment) from the FAS analysis of change at end of Period 2 from baseline in eGFR (MDRD).
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 87 | 44
fold change | 0.99 [0.98 to 1.01] | 1.01 [0.98 to 1.03]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 0.99, 90% CI 2-sided [0.96 to 1.02] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Adjusted Geometric Mean-Fold Change at End of Period 2 From End of Period 1 in eGFR Using MDRD
Description: eGFR was calculated using the MDRD equation with eGFR values normalized to 1.73 m^2 body surface area.
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS (OC); three participants were excluded (took wrong treatment) from the FAS analysis of change at end of Period 2 from end of Period 1 in eGFR (MDRD).
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 87 | 44
fold change | 1.04 [1.02 to 1.06] | 1.00 [0.97 to 1.03]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 1.04, 90% CI 2-sided [1.00 to 1.08] — ANCOVA with change in logarithmic eGFR (MDRD) from Period 2 baseline/end of Period 1 as dependent variable, treatment and logarithmic Period 2 baseline/end of Period 1 as covariate

7. Secondary Outcome: Adjusted Geometric Mean-Fold Change at End of Period 1 From Baseline in eGFR Using the Cockcroft-Gault Equation
Description: eGFR was calculated using the Cockcroft-Gault equation normalized to 1.73 m^2 body surface area. Baseline was defined as the mean of the values obtained at Screening and on predose in Period 1/Day 1.
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS OC; one participant was excluded (took wrong treatment) from the FAS analysis of change at end of Period 1 from baseline in eGFR (Cockcroft-Gault).
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 92 | 46
fold change | 0.96 [0.95 to 0.98] | 1.01 [0.99 to 1.04]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 0.95, 90% CI 2-sided [0.92 to 0.98] — ANCOVA with change in logarithmic eGFR (Cockcroft-Gault) from baseline as dependent variable, treatment and logarithmic baseline as covariate

8. Secondary Outcome: Adjusted Geometric Mean-Fold Change at End of Period 2 From Baseline in eGFR Using the Cockcroft-Gault Equation
Description: as for outcome 7
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS OC; three participants were excluded (took wrong treatment) from the FAS analysis of change at end of Period 2 from baseline in eGFR (Cockcroft-Gault).
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 87 | 44
fold change | 1.00 [0.98 to 1.01] | 1.01 [0.98 to 1.03]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 0.99, 90% CI 2-sided [0.97 to 1.02] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Adjusted Geometric Mean-Fold Change at End of Period 2 From End of Period 1 in eGFR Using the Cockcroft-Gault Equation
Description: eGFR was calculated using the Cockcroft-Gault equation normalized to 1.73 m^2 body surface area.
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS OC; three participants were excluded (took wrong treatment) from the FAS analysis of change at end of Period 2 from end of Period 1 in eGFR (Cockcroft-Gault).
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 87 | 44
fold change | 1.03 [1.01 to 1.05] | 1.00 [0.97 to 1.02]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 1.04, 90% CI 2-sided [1.01 to 1.07] — ANCOVA with change in logarithmic eGFR (Cockcroft-Gault) from Period 2 baseline/end of Period 1 as dependent variable, treatment and logarithmic Period 2 baseline/end of Period 1 as covariate

10. Secondary Outcome: Adjusted Geometric Mean-Fold Change at End of Period 1 From Baseline in Serum Creatinine
Description: Blood samples were collected from participants at screening, predose on Day 1 of Period 1, on the last day of Period 1 and on the last day of Period 2 for assessment of serum creatinine levels. Serum creatinine values in milligrams per deciliter (mg/dL) reported by the central laboratory were used. Baseline for serum creatinine was defined as the mean of values obtained at screening and predose on Day 1 of Period 1.
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS OC; one participant was excluded (took wrong treatment) from the FAS analysis of change at end of Period 1 from baseline in serum creatinine.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 92 | 46
fold change | 1.04 [1.02 to 1.06] | 0.99 [0.97 to 1.01]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 1.05, 90% CI 2-sided [1.02 to 1.08] — ANCOVA with change in logarithmic creatinine from baseline as dependent variable, treatment and logarithmic baseline as covariate

11. Secondary Outcome: Adjusted Geometric Mean-Fold Change From End of Period 2 From Baseline in Serum Creatinine
Description: Blood samples were collected from participants at screening, predose on Day 1 of Period 1, on the last day of Period 1 and on the last day of Period 2 for assessment of serum creatinine levels. Serum creatinine values in mg/dL reported by the central laboratory were used. Baseline for serum creatinine was defined as the mean of values obtained at screening and predose on Day 1 of Period 1.
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS OC; three participants were excluded (took wrong treatment) from the FAS analysis of change at end of Period 2 from baseline in serum creatinine.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 87 | 44
fold change | 1.00 [0.99 to 1.02] | 1.00 [0.97 to 1.02]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 1.01, 90% CI 2-sided [0.98 to 1.04] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Adjusted Geometric Mean-Fold Change at End of Period 2 From End of Period 1 in Serum Creatinine
Description: Blood samples were collected from participants at screening, predose on Day 1 of Period 1, on the last day of Period 1 and on the last day of Period 2 for assessment of serum creatinine levels. Serum creatinine values in mg/dL reported by the central laboratory were used.
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS OC; three participants were excluded (took wrong treatment) from the FAS analysis of change at end of Period 2 from end of Period 1 in serum creatinine.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 87 | 44
fold change | 0.97 [0.95 to 0.99] | 1.00 [0.98 to 1.03]
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Ratio of adjusted geometric mean-fold change (CP-690,550-placebo vs. placebo-placebo); Test type: Superiority or Other; ANCOVA; Ratio of Adjusted Geo Mean-Fold Change = 0.97, 90% CI 2-sided [0.94 to 1.00] — ANCOVA with change in logarithmic creatinine from Period 2 baseline/the end of Period 1 as dependent variable, treatment and Period 2 baseline/the end of Period 1 as covariate

13. Secondary Outcome: Percentage of Participants Achieving an American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: greater than or equal to (≥)20 percent (%) improvement in tender joint count; ≥20% improvement in swollen joint count; and ≥20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Day 1 of Period 1 to Day 43 of Period 1, Day 1 of Period 1 to Day 29 of Period 2
Population: FAS, missing values while participant was still enrolled utilized last observation carried forward (LOCF) imputation while participants with missing values after a participant was discontinued from study participation (for any reason) were considered to be nonresponders (nonresponder imputation [NRI])
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 97 | 51
percentage of participants
  End of Period 1 (Day 43) | 57.73 | 21.57
  End of Period 2 (Day 29) | 45.36 | 29.41
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Between-group difference in ACR20 Response at End of Period 1; Test type: Superiority or Other; p < 0.001, Normal approximation for proportions — Two-sided test at 5% significance level; Mean Difference (Final Values) = 36.16, 90% CI 2-sided [23.60 to 48.73], Standard Error of Mean 7.64
Statistical Analysis 2: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Between-group difference in ACR20 Response at End of Period 2; Test type: Superiority or Other; p = 0.050, Normal approximation for proportions — Two-sided test at 5% significance level; Mean Difference (Final Values) = 15.95, 90% CI 2-sided [2.56 to 29.34], Standard Error of Mean 8.14

14. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: ≥50% improvement in tender or swollen joint counts and 50% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a HAQ, and 5) CRP at each visit.
Time Frame: Day 1 of Period 1 to Day 43 of Period 1, Day 1 of Period 1 to Day 29 of Period 2
Population: FAS (NRI, LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 97 | 51
percentage of participants
  End of Period 1 (Day 43) | 28.87 | 7.84
  End of Period 2 (Day 29) | 26.80 | 9.80
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Between-group difference in ACR50 Response at End of Period 1; Test type: Superiority or Other; p < 0.001, Normal approximation for proportions — Two-sided test at 5% significance level; Mean Difference (Final Values) = 21.02, 90% CI 2-sided [11.24 to 30.80], Standard Error of Mean 5.94
Statistical Analysis 2: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Between-group difference in ACR50 Response at End of Period 2; Test type: Superiority or Other; p = 0.006, Normal approximation for proportions — Two-sided test at 5% significance level; Mean Difference (Final Values) = 17.00, 90% CI 2-sided [6.92 to 27.08], Standard Error of Mean 6.13

15. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: ≥70% improvement in tender or swollen joint counts and 70% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant' assessment of functional disability via a HAQ, and 5) CRP at each visit.
Time Frame: Day 1 of Period 1 to Day 43 of Period 1, Day 1 of Period 1 to Day 29 of Period 2
Population: FAS (NRI, LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 97 | 51
percentage of participants
  End of Period 1 (Day 43) | 18.56 | 0.00
  End of Period 2 (Day 29) | 9.28 | 1.96
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Between-group difference in ACR70 Response at End of Period 1; Test type: Superiority or Other; p < 0.001, Normal approximation for proportions — Two-sided test at 5% significance level; Mean Difference (Final Values) = 18.56, 90% CI 2-sided [12.06 to 25.05], Standard Error of Mean 3.95
Statistical Analysis 2: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Between-group difference in ACR70 Response at End of Period 2; Test type: Superiority or Other; p = 0.038, Normal approximation for proportions — Two-sided test at 5% significance level; Mean Difference (Final Values) = 7.32, 90% CI 2-sided [1.51 to 13.12], Standard Error of Mean 3.53

16. Secondary Outcome: Least Squares (LS) Mean Change at End of Period 1 From Baseline in Disease Activity Score Based on 28-Joint Count CRP (DAS28-3 [CRP])
Description: DAS28 calculated from the tender/painful joint count, swollen joint count (SJC) using the 28 joints count, and CRP value. DAS28 less than or equal to (≤)3.2 equals (=) low disease activity, DAS28 greater than (>)3.2 to 5.1 = moderate to high disease activity.
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 93 | 45
score on a scale | -1.71 (0.13) | -0.55 (0.19)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -1.16, 90% CI 2-sided [-1.53 to -0.78], Standard Error of Mean 0.23 — Linear mixed-effects model for longitudinal data was used with actual value as dependent variable, treatment group, visit (baseline, end of Period 1, end of Period 2), treatment group by visit interaction as fixed effect, participant as random effect

17. Secondary Outcome: LS Mean Change at End of Period 2 From Baseline in DAS28-3 (CRP)
Description: DAS28 calculated from the tender/painful joint count, SJC using the 28 joints count, and CRP value. DAS28 ≤3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 44
score on a scale | -1.36 (0.12) | -0.89 (0.17)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.028, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -0.47, 90% CI 2-sided [-0.83 to -0.12], Standard Error of Mean 0.21 — [estimate comment as in outcome 16, analysis 1]

18. Secondary Outcome: LS Mean Change at End of Period 2 From End of Period 1 in DAS28-3 (CRP)
Description: as for outcome 17
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 43
score on a scale | 0.35 (0.12) | -0.34 (0.18)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = 0.68, 90% CI 2-sided [0.32 to 1.04], Standard Error of Mean 0.22 — [estimate comment as in outcome 16, analysis 1]

19. Secondary Outcome: LS Mean Change at End of Period 1 From Baseline DAS28-4 (CRP)
Description: DAS28 calculated from the number of SJC and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 ≤3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 93 | 44
score on a scale | -1.88 (0.14) | -0.62 (0.21)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -1.26, 90% CI 2-sided [-1.67 to -0.84], Standard Error of Mean 0.25 — [estimate comment as in outcome 16, analysis 1]

20. Secondary Outcome: LS Mean Change at End of Period 2 From Baseline DAS28-4 (CRP)
Description: DAS28 calculated from the number of SJC and PJC using the 28 joints count, the ESR (mm/hour) and PGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 ≤3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 44
score on a scale | -1.46 (0.13) | -0.96 (0.19)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.031, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -0.50, 90% CI 2-sided [-0.88 to -0.12], Standard Error of Mean 0.23 — [estimate comment as in outcome 16, analysis 1]

21. Secondary Outcome: LS Mean Change at End of Period 2 From End of Period 1 DAS28-4 (CRP)
Description: as for outcome 20
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 42
score on a scale | 0.42 (0.14) | -0.34 (0.20)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = 0.76, 90% CI 2-sided [0.36 to 1.15], Standard Error of Mean 0.24 — [estimate comment as in outcome 16, analysis 1]

22. Secondary Outcome: LS Mean Change at End of Period 1 From Baseline in Tender/Painful Joint Count
Description: 68 joints were assessed by a joint assessor to determine the number of joints that were considered tender or painful Assessed joints included: upper body (temporomandibular, sternoclavicular, acromioclavicular), upper extremity (shoulder, elbow, wrist, MCP, thumb interphalangeal [IP], PIP, and distal interphalangeals [DIP]), and lower extremity (hip, knee, ankle, tarsus, metatarsophalangeals [MTP], great toe IP, proximal and distal interphalangeals combined [PIP]).
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: tender/painful joints
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 93 | 45
tender/painful joints | -9.88 (1.16) | -5.79 (1.66)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -4.09, 90% CI 2-sided [-7.44 to -0.74], Standard Error of Mean 2.02 — [estimate comment as in outcome 16, analysis 1]

23. Secondary Outcome: LS Mean Change at End of Period 2 From Baseline in Tender/Painful Joint Count
Description: 68 joints were assessed by a joint assessor to determine the number of joints that were considered tender or painful Assessed joints included: upper body (temporomandibular, sternoclavicular, acromioclavicular), upper extremity (shoulder, elbow, wrist, MCP, thumb IP, PIP, and DIP), and lower extremity (hip, knee, ankle, tarsus, MTP, great toe IP, proximal and distal interphalangeals combined [PIP]).
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: tender/painful joints
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 45
tender/painful joints | -8.13 (1.02) | -8.27 (1.44)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.936, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = 0.14, 90% CI 2-sided [-2.78 to 3.06], Standard Error of Mean 1.76 — [estimate comment as in outcome 16, analysis 1]

24. Secondary Outcome: LS Mean Change at End of Period 2 From End of Period 1 in Tender/Painful Joint Count
Description: as for outcome 23
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: tender/painful joints
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 44
tender/painful joints | 1.75 (1.11) | -2.48 (1.58)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = 4.23, 90% CI 2-sided [1.04 to 7.42], Standard Error of Mean 1.93 — [estimate comment as in outcome 16, analysis 1]

25. Secondary Outcome: LS Mean Change at End of Period 1 From Baseline in Swollen Joint Count
Description: Swollen joint count included 66 joints. Assessor assessed joints for swelling using the following scale: present/absent/not done/not applicable (to be used for artificial joints). Joints assessed included: upper body (temporomandibular, sternoclavicular, acromioclavicular), upper extremity (shoulder, elbow, wrist, MCP, thumb IP, PIP, and DIP), and lower extremity (knee, ankle, tarsus, MTP, great toe IP, proximal and distal interphalangeals combined [PIP]).
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 93 | 45
swollen joints | -7.07 (0.59) | -4.81 (0.84)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -2.26, 90% CI 2-sided [-3.96 to -0.55], Standard Error of Mean 1.03 — [estimate comment as in outcome 16, analysis 1]

26. Secondary Outcome: LS Mean Change at End of Period 2 From Baseline in Swollen Joint Count
Description: as for outcome 25
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 45
swollen joints | -6.63 (0.64) | -5.83 (0.91)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.472, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -0.80, 90% CI 2-sided [-2.64 to 1.04], Standard Error of Mean 1.11 — [estimate comment as in outcome 16, analysis 1]

27. Secondary Outcome: LS Mean Change at End of Period 2 From End of Period 1 in Swollen Joint Count
Description: as for outcome 25
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 44
swollen joints | 0.43 (0.59) | -1.02 (0.84)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.158, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = 1.46, 90% CI 2-sided [-0.24 to 3.15], Standard Error of Mean 1.03 — [estimate comment as in outcome 16, analysis 1]

28. Secondary Outcome: LS Mean Change at End of Period 1 From Baseline in CRP
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 93 | 46
mg/L | -13.81 (2.17) | -0.08 (3.01)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -13.73, 90% CI 2-sided [-19.87 to -7.59], Standard Error of Mean 3.71 — [estimate comment as in outcome 16, analysis 1]

29. Secondary Outcome: LS Mean Change at End of Period 2 From Baseline in CRP
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 44
mg/L | -8.37 (2.34) | 0.53 (3.29)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -8.89, 90% CI 2-sided [-15.58 to -2.21], Standard Error of Mean 4.04 — [estimate comment as in outcome 16, analysis 1]

30. Secondary Outcome: LS Mean Change at End of Period 2 From End of Period 1 in CRP
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 44
mg/L | 5.44 (1.71) | 0.61 (2.44)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.107, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = 4.84, 90% CI 2-sided [-0.10 to 9.77], Standard Error of Mean 2.98 — [estimate comment as in outcome 16, analysis 1]

31. Secondary Outcome: LS Mean Change at End of Period 1 From Baseline in Patient Global Assessment of Arthritis (PGAA)
Description: Participants answered the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 millimeter (mm) visual analog scale (VAS), where 0 mm = very well and 100 mm = very poorly.
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 93 | 45
mm | -23.28 (2.81) | -7.38 (3.98)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -15.90, 90% CI 2-sided [-23.96 to -7.84], Standard Error of Mean 4.87 — [estimate comment as in outcome 16, analysis 1]

32. Secondary Outcome: LS Mean Change at End of Period 2 From Baseline in PGAA
Description: Participants answered the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" The participants responses were recorded using a 100 mm VAS, where 0 mm = very well and 100 mm = very poorly.
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 45
mm | -16.12 (2.87) | -10.41 (4.03)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.251, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -5.70, 90% CI 2-sided [-13.90 to 2.50], Standard Error of Mean 4.95 — [estimate comment as in outcome 16, analysis 1]

33. Secondary Outcome: LS Mean Change at End of Period 2 From End of Period 1 in PGAA
Description: as for outcome 32
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 44
mm | 7.16 (2.54) | -3.03 (3.62)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = 10.19, 90% CI 2-sided [2.87 to 17.52], Standard Error of Mean 4.42 — [estimate comment as in outcome 16, analysis 1]

34. Secondary Outcome: LS Mean Change at End of Period 1 From Baseline in Physician Global Assessment of Arthritis
Description: A physician assessed how the participant's overall arthritis appeared at the time of the visit. This was an evaluation based on the participant's disease signs, functional capacity and physical examination. The physician's response was recorded using a 100 mm VAS, where 0 mm = very good and 100 mm = very poor.
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 93 | 45
mm | -29.83 (2.24) | -14.71 (3.19)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -15.12, 90% CI 2-sided [-21.58 to -8.67], Standard Error of Mean 3.90 — [estimate comment as in outcome 16, analysis 1]

35. Secondary Outcome: LS Mean Change at End of Period 2 From Baseline in Physician Global Assessment of Arthritis
Description: as for outcome 34
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 45
mm | -24.61 (2.76) | -22.21 (3.89)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.616, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -2.40, 90% CI 2-sided [-10.30 to 5.50], Standard Error of Mean 4.77 — [estimate comment as in outcome 16, analysis 1]

36. Secondary Outcome: LS Mean Change at End of Period 2 From End of Period 1 in Physician Global Assessment of Arthritis
Description: as for outcome 34
Time Frame: Day 43 of Period 1, Day 29 of Period 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 44
mm | 5.22 (2.39) | -7.50 (3.41)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = 12.72, 90% CI 2-sided [5.82 to 19.62], Standard Error of Mean 4.17 — [estimate comment as in outcome 16, analysis 1]

37. Secondary Outcome: LS Mean Change at End of Period 1 From Baseline in Patient Assessment of Arthritis Pain
Description: Participant's assessed the severity of their arthritis pain using a 100 mm VAS placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponded to the magnitude of their pain.
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 93 | 46
mm | -23.53 (2.61) | -8.23 (3.69)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -15.30, 90% CI 2-sided [-22.78 to -7.82], Standard Error of Mean 4.52 — [estimate comment as in outcome 16, analysis 1]

38. Secondary Outcome: LS Mean Change at End of Period 2 From Baseline in Patient Assessment of Arthritis Pain
Description: as for outcome 37
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 45
mm | -14.70 (2.80) | -9.08 (3.94)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.247, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -5.62, 90% CI 2-sided [-13.62 to 2.38], Standard Error of Mean 4.83 — [estimate comment as in outcome 16, analysis 1]

39. Secondary Outcome: LS Mean Change at End of Period 2 From End of Period 1 in Patient Assessment of Arthritis Pain
Description: as for outcome 37
Time Frame: Day 43 of Period 2, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 45
mm | 8.83 (2.69) | -0.85 (3.81)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.040, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = 9.68, 90% CI 2-sided [1.95 to 17.41], Standard Error of Mean 4.67 — [estimate comment as in outcome 16, analysis 1]

40. Secondary Outcome: LS Mean Change at End of Period 1 From Baseline Health Assessment Questionnaire Disability Index (HAQ-DI) Score
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Day 1 of Period 1, Day 43 of Period 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 93 | 46
score on a scale | -0.44 (0.06) | -0.04 (0.08)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -0.39, 90% CI 2-sided [-0.56 to -0.23], Standard Error of Mean 0.10 — [estimate comment as in outcome 16, analysis 1]

41. Secondary Outcome: LS Mean Change at End of Period 2 From Baseline HAQ-DI Score
Description: as for outcome 40
Time Frame: Day 1 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 45
score on a scale | -0.34 (0.05) | -0.17 (0.07)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.053, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = -0.17, 90% CI 2-sided [-0.31 to -0.03], Standard Error of Mean 0.09 — [estimate comment as in outcome 16, analysis 1]

42. Secondary Outcome: LS Mean Change at End of Period 2 From End of Period 1 HAQ-DI Score
Description: as for outcome 40
Time Frame: Day 43 of Period 1, Day 29 of Period 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Number analyzed (Participants) | 90 | 45
score on a scale | 0.09 (0.04) | -0.13 (0.06)
Statistical Analysis 1: Comparison: CP-690,550/Placebo vs Placebo/Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — Two-sided test at 5% significance level; Mean Difference (Final Values) = 0.22, 90% CI 2-sided [0.10 to 0.35], Standard Error of Mean 0.07 — [estimate comment as in outcome 16, analysis 1]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550/Placebo | Placebo/Placebo
Serious Adverse Events (participants affected / at risk) | 2/97 | 0/51
Other Adverse Events (participants affected / at risk) | 32/97 | 26/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550/Placebo (N=97) | Placebo/Placebo (N=51)
Bronchopneumonia (Infections and infestations) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550/Placebo (N=97) | Placebo/Placebo (N=51)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Medical device complication (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 8 | 3
Oral herpes (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 2 | 0
Blood urea increased (Investigations) | 0 | 1
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.